CLINICAL TRIAL: NCT00609986
Title: Intravenous Insulin Protocol in Diabetes and Renal Transplantation Study
Brief Title: IV Insulin Protocol in Diabetes and Renal Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Kathie Hermayer, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR #17383; ADA 7-07-CR-22
Record Dates: First submitted 2008-01-02; First posted 2008-02-07 (Estimated); Results first posted 2013-08-07 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-08

CONDITIONS: Kidney Transplantation; Diabetes; Hyperglycemia
Keywords: Kidney; Transplantation; Diabetes; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia | interventions — Insulin; Insulin, Isophane; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive (Experimental): The experimental group will receive the intravenous regular insulin infusion protocol for the maintenance of blood sugar levels 70-110 mg/dL while hospitalized up to 7 am post operative day #3 and after hospitalization will receive subcutaneous insulin to maintain blood sugar levels 70-140 mg/dL.
  Interventions: Drug: insulin
- Control (Active Comparator): The control group will receive subcutaneous insulin injections (NPH or glargine and aspartame) to maintain a blood sugar level between 70-180 mg/dL while hospitalized and after hospitalization subcutaneous insulin to maintain blood sugar levels 90-180 mg/dL.
  Interventions: Drug: NPH Insulin or glargine insulin and aspartame insulin

INTERVENTIONS:
Drug: insulin — The intravenous regular insulin infusion will be delivered continuously during the transplant surgery and after surgery for a total of three days. While receiving the insulin infusion, the dose will be calculated to keep the blood sugar levels between 70-110 mg/dL.
  After the regular insulin infusion is discontinued, the blood sugar levels will be measured by a finger stick blood glucose up to 5-6 times per day and the blood sugar levels will be corrected by a subcutaneous basal-bolus insulin injection for a blood sugar goal 70-110 mg/dL.
  Upon discharge from the hospital, the patient will be placed on a basal-bolus regimen consisting of 3-4 insulin injections to maintain a blood sugar between 70-140.
  Arms: Intensive
Drug: NPH Insulin or glargine insulin and aspartame insulin — The NPH or glargine and aspartame insulin will be given subcutaneously using a small-short needle to administer the insulin.
  The blood sugar level will be checked every 1 hour while in the operating room and treated with rapid-acting insulin as needed to keep the blood sugar levels 70-180 mg/dL. The blood sugar level will be checked every 4 hours when in the recovery room and on the 6 East transplant unit. Once the patient is able to eat, the blood sugar will be checked five times a day (before meals, at bedtime, and at 3:00 am). Long-acting and rapid-acting insulin will be used to maintain the target blood sugar level.
  Upon discharge from the hospital, the patient will be placed on a minimum of one to two insulin injections to maintain a blood sugar between 90-180 mg/dL
  Arms: Control

SUMMARY:
Purpose: The purpose of this study is to provide tight blood sugar control using insulin given through the veins at the time of kidney transplantation and up to 3 days after surgery. After release from the hospital, the patient will control blood sugar with subcutaneous insulin injections or pills. With this approach, outcomes should improve for diabetic transplant patients such as longer life of the new kidney, fewer hospital readmissions, decreased associated infections, and other advantages.

Hypothesis: It is hypothesized that intensive glycemic control will lead to better clinical and biochemical outcomes and improved long-term graft survival.

DETAILED DESCRIPTION:
Research Design: A randomized control trial comparing intensive intravenous insulin (IVI) for use in the hospital followed by intensive subcutaneous (sc) insulin use for in-patient and out-patient glycemic control will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and greater,
* Diabetes diagnosis (Type 1 and Type 2, awaiting a living or cadaveric renal transplant, renal transplant candidates admitted to MUSC medical center for a donor kidney, FBG >100 mg/dL per admission screening labs, random BG >120mg/dL per admission screening labs, and
* Willing and able to provide informed consent

Exclusion Criteria:

* History of an active GI bleed in the previous 3 mos,
* Scheduled to receive a simultaneous pancreas transplant,
* History of a functioning pancreatic transplant,
* Patient currently managed on an insulin pump,
* Unable or unwilling to provide informed consent, and
* Unable to commit to the study protocol including the outpatient follow-up phase of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2007-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathie L. Hermayer, MD, MS, Principal Investigator — Medical University of South Carolina, Division of Endocrinology
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Bellon F, Sola I, Gimenez-Perez G, Hernandez M, Metzendorf MI, Rubinat E, Mauricio D. Perioperative glycaemic control for people with diabetes undergoing surgery. Cochrane Database Syst Rev. 2023 Aug 1;8(8):CD007315. doi: 10.1002/14651858.CD007315.pub3. PMID 37526194
- [Derived] Lo C, Toyama T, Oshima M, Jun M, Chin KL, Hawley CM, Zoungas S. Glucose-lowering agents for treating pre-existing and new-onset diabetes in kidney transplant recipients. Cochrane Database Syst Rev. 2020 Jul 30;8(8):CD009966. doi: 10.1002/14651858.CD009966.pub3. PMID 32803882

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Medical University of South Carolina prior to receiving a renal transplant.
Period: Overall Study
Arm/Group | Intensive | Control
Started | 52 | 52
Received Transplant | 44 | 49
Completed | 44 | 49
Not Completed | 8 | 3
Not completed — Did not receive transplant or treatment | 8 | 3

BASELINE CHARACTERISTICS:
Population: The intent-to-treat anaylsis consisted only of the 93 participants that underwent a renal transplant.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive | Control | Total
Number analyzed (Participants) | 44 | 49 | 93
Age Continuous [Mean (Standard Deviation); unit: years] | 58 (9.8) | 56.3 (9.6) | 57.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 30 | 35 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 28 | 56
  White | 15 | 18 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Delayed Graft Function
Description: Need for dialysis in the first week post-transplant in a patient who required dialysis pre-transplantation or day-10 post-transplant creatinine concentration above 2.5 mg/dl.
Time Frame: 10 days
Population: The intent-to-treat analysis set consisted of the participants that underwent a renal transplant.
Measure: Number; unit: participants
Arm/Group | Intensive | Control
Number analyzed (Participants) | 44 | 49
participants | 8 | 12

2. Secondary Outcome: Severe Hypoglycemia
Description: Blood glucose less than 40 mg/dl
Time Frame: 30 months
Population: The intent-to-treat analysis set consisted of the participants that underwent a renal transplant.
Measure: Number; unit: participants
Arm/Group | Intensive | Control
Number analyzed (Participants) | 44 | 49
participants | 7 | 2

3. Primary Outcome: Acute/Active Rejection
Description: Grades IA through III and antibody immediate rejection, either A (immediate or hyperacute) or B (delayed or accelerated acute) were diagnosed and classified based on renal allograft biopsies according to the Banff 97 Working Classification of Renal Allograph Pathology.
Time Frame: 30 months
Population: The intent-to-treat analysis set consisted of the participants that underwent a renal transplant.
Measure: Number; unit: participants
Arm/Group | Intensive | Control
Number analyzed (Participants) | 44 | 49
participants | 9 | 2

4. Secondary Outcome: Severe Hyperglycemia
Description: Blood glucose greater than 350 mg/dl.
Time Frame: 30 months
Population: The intent-to-treat analysis set consisted of the participants that underwent a renal transplant.
Measure: Number; unit: participants
Arm/Group | Intensive | Control
Number analyzed (Participants) | 44 | 49
participants | 5 | 12

ADVERSE EVENTS:
Arm/Group | Intensive | Control
Serious Adverse Events (participants affected / at risk) | 0/44 | 1/49
Other Adverse Events (participants affected / at risk) | 12/44 | 14/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive (N=44) | Control (N=49)
renal graft thrombosis (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive (N=44) | Control (N=49)
severe hypoglycemia (Endocrine disorders) | 7 (8) | 2 (2)
severe hyperglycemia (Endocrine disorders) | 5 (5) | 12 (25)

LIMITATIONS AND CAVEATS:
A limitation of the trial was that the majority of the patients enrolled in the study were African American, and therefore the findings cannot be extended to groups of other ethnic groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No